CLINICAL TRIAL: NCT03150160
Title: A 6-week, Double Masked, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Twice-daily Brinzolamide 1%/Brimonidine 0.2% Fixed Dose Combination as an Adjunctive Therapy to Travoprost 0.004% in Reducing Intraocular Pressure in Patients With Normal Tension Glaucoma
Brief Title: Additive Effect of Twice-daily Brinzolamide 1%/Brimonidine 0.2%Combination as an Adjunctive Therapy to Travoprost in Patients With Normal Tension Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVJ499A2404
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-10

CONDITIONS: Glaucoma
Keywords: travoprost; brinzolamide 1%/brimonidine 0.2%; normal tension glaucoma; intraocular pressure; efficacy; safety
MeSH Terms: conditions — Glaucoma; Low Tension Glaucoma | interventions — brinzolamide; Brimonidine Tartrate; Travoprost; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This was a multicenter, randomized, double-masked, two-arm, placebo-controlled, parallel group study in patients with normal tension glaucoma who were insufficiently controlled on travoprost 0.004% (Travatan) monotherapy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simbrinza + Travatan (Experimental): Brinzolamide 1%/brimonidine 0.2% fixed combination + travoprost 0.004% ophthalmic solution
  Interventions: Drug: brinzolamide 1%/brimonidine 0.2% fixed combination; Drug: travoprost 0.004% ophthalmic solution
- Placebo + Travatan (Placebo Comparator): Placebo + travoprost 0.004% ophthalmic solution
  Interventions: Drug: Placebo; Drug: travoprost 0.004% ophthalmic solution

INTERVENTIONS:
Drug: brinzolamide 1%/brimonidine 0.2% fixed combination — One drop applied topically to the affected eye(s) in the morning and evening
  Other Names: Simbrinza
  Arms: Simbrinza + Travatan
Drug: Placebo — One drop applied topically to the affected eye(s) in the morning and evening
  Arms: Placebo + Travatan
Drug: travoprost 0.004% ophthalmic solution — One drop applied topically to the affected eye(s) in the evening
  Other Names: Travatan

SUMMARY:
The purpose of this study was to determine the incremental intraocular pressure (IOP) lowering that is achieved when Simbrinza is used adjunctively to Travatan in patients with normal tension glaucoma that may benefit from further IOP lowering.

DETAILED DESCRIPTION:
This study was prematurely terminated due to administrative reasons and not due to any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent
* Diagnosed with normal tension glaucoma
* Intraocular pressure measurements in at least 1 eye as specified in the protocol
* Willing and able to attend all study visits

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs
* Use of medications prohibited by the protocol
* Pregnant or nursing
* Of child-bearing potential unless using contraception, as specified in the protocol
* Any form of glaucoma other than open angle glaucoma in either eye
* Chronic, recurrent or severe inflammatory eye disease
* Ocular trauma or surgery within the past 6 months in either eye; ocular infection or laser surgery within the past 3 months in either eye (all from screening)
* Conditions which would make the patient, in the opinion of the Investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized patients (1). Note: No patients were randomized to the Simbrinza + Travatan arm.
Groups:
- Simbrinza + Travatan: Brinzolamide 1%/brimonidine 0.2% fixed combination (morning and evening) + travoprost 0.004% ophthalmic solution (evening)
- Placebo + Travatan: Placebo (morning and evening) + travoprost 0.004% ophthalmic solution (evening)
Period: Overall Study
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the Simbrinza + Travatan arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simbrinza + Travatan | Placebo + Travatan | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Diurnal IOP at Week 6
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry in millimeters mercury (mmHg). Diurnal IOP was defined as the average of the 9:00 am and 11:00 am time points. A more negative change value indicates a greater amount of improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: At the time of the premature termination of this study, only 1 patient was randomized. Therefore, the planned efficacy and safety analyses could not be performed. No data to report.
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in IOP at Week 6
Description: IOP was measured by Goldmann applanation tonometry in mmHg. A more negative percent change value indicates a greater amount of improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Diurnal IOP at Week 6
Description: IOP was measured by Goldmann applanation tonometry in mmHg. Diurnal IOP was defined as the average of the 9:00 and 11:00 time points. One (study eye) contributed to the analysis.
Time Frame: Week 6
Population: as for outcome 1
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Baseline in IOP for Each Time Point at Week 6
Description: IOP was measured by Goldmann applanation tonometry in mmHg. A more negative change value indicates a greater amount of improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (9:00 am and 11:00 am), Week 6 (9:00 am and 11:00 am)
Population: as for outcome 1
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage Change From Baseline in IOP for Each Time Point at Week 6
Description: as for outcome 2
Time Frame: Baseline, Week 6
Population: as for outcome 1
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately six weeks.
Description: The Safety analysis set included all patients exposed to at least one dose of any study therapy. Note: Number at risk for Simbrinza + Travatan is reported as 0 because no patients were exposed to this study therapy.
Arm/Group | Simbrinza + Travatan | Placebo + Travatan
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simbrinza + Travatan (N=0) | Placebo + Travatan (N=1)
common cold (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03150160/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03150160/SAP_001.pdf